CLINICAL TRIAL: NCT01087255
Title: Caregivers and Internet Based Monitoring to Improve Medication Use in HPHC Enrollees With Chronic Kidney Disease
Brief Title: Caregivers and Electronic Medication Monitoring in Chronic Kidney Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harvard Pilgrim Health Care (Other)
Responsible Party: Connie Mah Trinacty, PhD, Assistant Professor, Department of Population Medicine, Harvard Pilgrim Health Care Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PF000123
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2010-03

CONDITIONS: Chronic Kidney Disease; Medication Adherence
Keywords: Caregiver-based interventions; Chronic Kidney Disease; Medication Adherence
MeSH Terms: conditions — Renal Insufficiency, Chronic; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Usual care patients will have outpatient care and monitoring procedures, as determined by them and their health care providers.
- Electronic Pillbox Monitoring System (Experimental): Usual care plus receive use of the wireless electronic pillbox and medication monitoring system
  Interventions: Device: Electronic Pillbox Monitoring System

INTERVENTIONS:
Device: Electronic Pillbox Monitoring System — Daily exposure for six months
  Other Names: MedMinder
  Arms: Electronic Pillbox Monitoring System

SUMMARY:
The objective of this pilot study is to explore barriers to medication adherence among HPHC members with CKD, particularly those not yet on dialysis, and to assess the feasibility and acceptability of a wireless, internet-based MedMinder system intervention among HPHC enrollees with CKD and their care partners. The investigators hypothesize that the intervention will improve medication use and adherence among patient members with CKD on complex medication treatment, and improve informal caregivers' ability to provide support for improved medication use among patient members.

DETAILED DESCRIPTION:
Adherence to medications is critical in managing chronic disease, yet it remains an issue across chronic conditions. Poor medication adherence leads to deteriorating health and subsequently to increased costs as a result of higher hospitalizations rates. Medication adherence in chronic kidney disease (CKD) is especially important because successful treatment can slow the progression to end-stage renal disease (ESRD), yet little research has focused on adherence in patients with early CKD. Numerous barriers to medication adherence exist, including the prescription of complex medication regimens, the often asymptomatic nature of early CKD, and the lack of social support for treatment adherence. While technology and support-based interventions show promise, there currently is no gold-standard approach to improving medication adherence. Thus, it is essential to pursue novel interventions that address barriers for patients with CKD to improve medication adherence and slow the progression to ESRD.

The long-range goal of this application is to improve medication adherence in chronic illness through the development of effective interventions that capitalize on patients' medication-taking context. The objective of this application, which is the next step to achieving that goal, is to pilot test the impact and acceptability of the MedMinder, a pillbox device that transmits medication-taking data via a secure internet-interface to patients, family members, and care managers, in a group of adult, Harvard Pilgrim Health Care (HPHC) members with CKD. To achieve this objective, in partnership with HPHC, we will recruit 120 members with diagnosed CKD stage III or IV to participate in a 6-month pre-post randomized-controlled trial. Participants will be randomized to either receive use of the MedMinder over a six-month period with access to telephone care management, or receive usual care of regular pillboxes with access to telephone care management.

Our primary aim is to test the feasibility and acceptability of the MedMinder intervention. The main components of the intervention include: (1) a plastic weekly pill box with programmable visual and auditory cues to prompt medication use, (2) generation of missed-dose alerts that can be sent via email, text message, or telephone to patients, family members, and HPHC care managers, (3) a secure internet site that permits customization of alerts and has graphical representations of medication use, and (4) aggregate adherence reports available to CKD care managers for patients who are participating in HPHC care management.

Our secondary aim is to assess the impact and acceptability of family and friend involvement in CKD member medication taking. We will document family and friend activities related to medication taking, the acceptability of family and friend involvement in member medication taking, and the impact such involvement has on medication use.

Findings of this proposed project would provide information on the feasibility of a technology-based adherence intervention, with medication-taking support, in patients with chronic disease. The results from this pilot will inform a future application for a more adequately powered study examining the intervention and measurement of structured support from others in medication taking.

ELIGIBILITY:
Inclusion Criteria:

* HPHC commercial- or Medicare-insured members with 2 or more distinct outpatient nephrology chronic kidney disease stage (CKD) III, IV, or V diagnoses in a 6-month period.
* 18 years old or older at the time they are identified as having CKD.
* An average of two prescription medications dispensed per month in the prior 6-months.
* Residence in MA, ME, or NH
* Residence in an area with MedMinder-participating cellular coverage (includes most major cellular carriers)

Exclusion Criteria:

* Dialysis or dialysis-related complication medical service claims in 6-month period preceding study entry.
* Atrius Health member
* Serious mental illness or cognitive dysfunction medical service claim in 6-month period preceding study entry
* Primary language other than English
* Unable to use a pillbox
* Have no eligible caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
medication adherence | 6 months
  We will calculate the proportion of days over a six month follow up period. We will calculate quantity dispensed on all chronic prescriptions filled to measure the number of days a patient had chronic medications available during the study period ("days covered"). Patients who switch treatment from one medication to another within the same therapeutic category will count toward adherence. Adherence is indicated by patients using >80% of prescribed doses.

CONTACTS AND LOCATIONS:
Overall Officials: Connie M Trinacty, PhD, Principal Investigator — Harvard Medical School and Harvard Pilgrim Health Care Institute; Ashley J Beard, PhD, Study Director — University of Michigan
Locations (1):
- Harvard Pilgrim Health Care, Wellesley, Massachusetts, United States